CLINICAL TRIAL: NCT00526032
Title: Melanoma Detection by Oblique-Incidence Optical Spectroscopy
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2006-0564
Record Dates: First submitted 2007-09-05; First posted 2007-09-06 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Skin Cancer
Keywords: Skin Cancer; Cancerous skin lesions; Melanoma Detection; Spectroscopic Oblique-Incidence Reflectometry; OIR Imaging Probe
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Spectroscopic Oblique-Incidence Reflectometry (OIR)
  Interventions: Procedure: OIR Imaging

INTERVENTIONS:
Procedure: OIR Imaging — Images from 4 different positions will be taken per lesion. The entire imaging procedure will take about 5 minutes per lesion.
  Other Names: imaging probe

SUMMARY:
Primary Objectives:

* To establish a statistically significant database: With Spectroscopic Oblique-Incidence Reflectometry (OIR) experimental system, we will obtain OIR spatio-spectral images of 1,000 human skin non-melanocytic and melanocytic lesions that, based on clinical diagnosis, are routinely biopsied and submitted for histopathologic diagnosis and of the adjacent normal skin for self-referencing. The experimental database will contain demographic information, clinical diagnoses, clinical images, OIR images, histopathologic diagnoses, and morphometric data on the lesions.
* To develop and validate a diagnostic algorithm:

  1. Classification: A subset (~50%) of OIR images collected will be used to complete the development of state-of-the-art image processing algorithms to extract robustly effective diagnostic features.
  2. Blind Testing and Evaluation: The algorithms established will be evaluated and validated in a prospective blind-test fashion using the complementary subset of the database that was not involved in designing the classifier. The sensitivity and specificity of the classification system will be evaluated based on the receiver-operating-characteristic (ROC) curve.
* To identify the pathophysiologic parameters responsible for the diagnostic optical features: The anatomic and physiologic sources of the diagnostic optical signatures will be identified by comparative analyses using the OIR images, microscopic histomorphometric techniques and theoretical modeling to test the following hypotheses:

  1. The calculated differences in hemoglobin oxygen saturation.
  2. Comparisons of the calculated size distributions of skin scattering centers with histologic and morphometric analyses of various cellular and tissue components of the skin lesions.
  3. The relative densities and distributions of the different anatomic and physiologic diagnostic features within the interrogation volumes are important diagnostic factors in OIR.

DETAILED DESCRIPTION:
The OIR imaging probe is designed to reflect light in a special way in order to take pictures of pigmented skin.

As part of your standard of care, your physician will check all skin lesions that may possibly be cancerous or pre-cancerous. Your physician will also check any non-cancerous lesions that are being removed for cosmetic reasons, such as warts and freckles.

If you agree to take part in this study, the study doctor will decide which lesions will be biopsied, as well as which lesions are eligible to be imaged. Pictures of the lesions (as well as healthy tissue nearby) will first be taken using a digital camera. The imaging probe and the area of the skin to be imaged will be cleaned with alcohol. After the imaging probe is placed over the lesion, a drop of baby oil will be applied to the skin. The imaging probe will then be lowered into contact with the skin, and the study staff will begin imaging. Twenty (20) images from 4 different positions will be taken per lesion.

Care will be taken to make sure that you cannot be identified from these images. For example, the study staff will avoid taking pictures of the face unless there are lesions there. After each lesion is imaged, the imaging device will be taken away and the skin surface cleaned. The entire imaging procedure, including preparation time, will take about 5 minutes per lesion.

Any hair on or around your lesions will be shaved or trimmed, if necessary. After all of the imaging is over, your lesion(s) will be biopsied. Your study doctor will decide which lesions require this kind of treatment as part of your standard care. Depending on what the study doctor decides, you will have either saucerization biopsies or excisional biopsies. A saucerization biopsy removes the entire lesion by cutting under it in a "scoop-like" manner. An excisional biopsy "cuts away" the entire lesion along with part of the surrounding skin.

A pathologist will receive your biopsied tissue and perform routine tests on the tissue. The test results will be available to the study doctor. Depending on whether the results are negative or positive, you may be informed of the results, as the biopsies are standard of care.

The images of your skin will be used for research to try to make the imaging probe more effective.

If you end your participation in this study early, your photographs and information will be removed from the researchers' database at that time. However, a record of your participation will remain in the database.

After all of the imaged lesions are biopsied, your participation in this study will be over.

This is an investigational study. The OIR imaging probe has not been approved by the FDA. Up to 1,000 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of any age, male or female, who are having a skin exam and are found to have a suspicious skin lesion on examination of their skin
2. Patients who agree to participate and sign the informed consent

Exclusion Criteria:

1. Patients who do not have a suspicious skin lesion
2. Patients who have not signed the informed consent and have agreed to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants having lesions on the skin that may be cancerous.
Sampling Method: Non-Probability Sample
Enrollment: 490 (Actual)
Dates: Start 2006-09; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Test OIR diagnostic medical tool (imaging probe) designed for early detection of skin cancers | 4 Years
  Observational study where patients getting skin biopsies of suspicious pigmented lesions were asked if their moles could be imaged with incidence optical spectroscopy. The light that was reflected back out was analyzed and hypothesized to differ from normal skin.

CONTACTS AND LOCATIONS:
Overall Officials: Madeleine Duvic, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org